CLINICAL TRIAL: NCT04216186
Title: Role of Coenzyme Q in Treatment of Attention Deficit Hyperactivity Disorder in Children
Brief Title: Role of Coenzyme Q in ADHD in Children
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: abeer salamah
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Atomoxetine Hydrochloride; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atomoxetine and Coenzyme Q (Active Comparator): Atomoxetine and Coenzyme Q
  Interventions: Drug: Atomoxetine; Drug: Coenzyme Q
- Placebo and Atomoxetine (Placebo Comparator): Placebo and Coenzyme Q
  Interventions: Drug: Coenzyme Q

INTERVENTIONS:
Drug: Atomoxetine — Atomoxetine once daily
  Other Names: atomox
  Arms: Atomoxetine and Coenzyme Q
Drug: Coenzyme Q — Coenzyme Q once daily

SUMMARY:
Role of Coenzyme Q in ADHD in Children

DETAILED DESCRIPTION:
Role of Coenzyme Q in ADHD in Children: will it add a benefit?

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADHD

Exclusion Criteria:

* Comorbidities like Autism, Anxiety, Obsessive compulsive disorder.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2030-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with improved CONNERS scale | 6 months
  The number of patients with improved CONNERS scale

CONTACTS AND LOCATIONS:
Overall Officials: Fatma G. Abdelkader, Msc, Principal Investigator — Pediatrics department - Kafr Elsheikh University; Osama A Elagamy, Prof., Principal Investigator — Pediatrics department - Kafr Elsheikh University; Abeer Salamah, Lecturer, Principal Investigator — Pediatrics department - Kafr Elsheikh University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gamal F, El Agami O, Salamah A. Coenzyme Q10 in the Treatment of Attention Deficit Hyperactivity Disorder in Children: A Randomized Controlled Trial. CNS Neurol Disord Drug Targets. 2022;21(8):717-723. doi: 10.2174/1871527320666211124093345. PMID 34819012